CLINICAL TRIAL: NCT01006954
Title: Comparison of Micro Dose Gonadotropin-Releasing Hormone (GnRH) Agonist Flare up & Flare Protocol in Poor Responders in Assisted Reproductive Technology (ART) Cycle
Brief Title: Outcome of Two Protocols in Poor Responders in Assisted Reproductive Technology (ART) Cycle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Emb-003
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2009-11

CONDITIONS: Infertility
Keywords: Poor responder; Flare up; Micro dose GnRH agonist flare up; IVF/ICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flare Up (Active Comparator): Flare up protocol in poor responders for IVF/ICSI
  Interventions: Drug: Flare up
- Microdose GnRh (Experimental): Microflare protocol in poor responders for IVF/ICSI
  Interventions: Drug: Microdose GnRh

INTERVENTIONS:
Drug: Microdose GnRh — Microflare protocol in poor responders for IVF/ICSI
  Other Names: Case
  Arms: Microdose GnRh
Drug: Flare up — Flare up protocol in poor responders for IVF/ICSI
  Other Names: Standard treatment
  Arms: Flare Up

SUMMARY:
About 9 to 24 % of women undergoing in vitro fertilization (IVF) treatment respond poorly to the usual gonadotrophin stimulation protocol applied. Several induction ovulation treatments have been suggested for increasing pregnancy rate. In this study, the investigators will compare the outcome of Microflare protocol and Flare up regimen in poor responders.

DETAILED DESCRIPTION:
In this randomized clinical trial study, a total of 200 infertile women with poor ovarian response who undergo IVF / ICSI treatment cycle at Royan Institute will enroll in this study and will randomly be divided into two groups of 100 patients. This study has been approved by Royan ethics committee and written consent will be obtained from each patient.

The patients will be randomized to one of two groups of Flare Up or Microdose GnRh agonist flare up.

Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), Estradiol, will be evaluated on day 2 or 3 and when follicle size become >14.

2 weeks after embryo transfer, the patients will be tested for serum β-hCG for assessing the pregnancy. The clinical pregnancy will be clarified by the number of women with gestational sacs on transvaginal sonography at 4-6 weeks of gestation. In the calculation of implantation, the number of gestational sacs will be considered.

ELIGIBILITY:
Inclusion Criteria:

Poor responders (Presence of at least two of following items is necessary for inclusion to the study)

* History of Cycle Cancellation
* History of oocyte number 3 (in previous cycle)
* History of Number of antral follicle < 5 in previous cycle
* Age≥38
* FSH>12 on day 2 or 3
* Ovarian Volume 3 cm3

Exclusion Criteria:

* Male factor (azospermi)
* Myoma ≥6cm
* One way ovary
* Tumor or cyst >13mm
* Age >42

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 12 months

SECONDARY OUTCOMES:
Cycle cancellation rates | 12 Months
Number of oocytes generated | 12 Months
Number of embryos generated | 12 Months
Implantation rate | 12 Months
Pregnancy rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tahereh Madani, MD, Study Chair — Royan Institute; Firoozeh Ghaffari, MD, Study Director — Royan Institute; Tahereh Madani, MD, Principal Investigator — Royan Institute
Locations (1):
- 1- Endocrinology and Female Infertility Department, Reproductive Medicine Research Centre, Royan Institute, ACECR, Tehran, Iran

REFERENCES:
- [Derived] Ghaffari F, Jahangiri N, Madani T, Khodabakhshi S, Chehrazi M. Randomized controlled trial of gonadotropin-releasing hormone agonist microdose flare-up versus flare-up among poor responders undergoing intracytoplasmic sperm injection. Int J Gynaecol Obstet. 2020 Jan;148(1):59-64. doi: 10.1002/ijgo.12988. Epub 2019 Oct 18. PMID 31569274
- See also: Related Info — http://WWW.Royaninstitute.org